CLINICAL TRIAL: NCT05578131
Title: The Effectiveness of Preoxygenation and Apneic Oxygenation Using High-flow Nasal Cannula for Pediatric Anesthetic Induction: a Prospective Randomized Open-label Clinical Trial
Brief Title: High-flow Nasal Cannula for Pediatric Anesthetic Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2209-089-1359
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia | interventions — Masks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal oxygen (Experimental)
  Interventions: Procedure: high flow nasal oxygen
- face mask (Active Comparator)
  Interventions: Procedure: face mask

INTERVENTIONS:
Procedure: high flow nasal oxygen — In the intervention group, pre-oxygenation was provided using HFNO via Optiflow THRIVE™ (Fisher and Paykel Healthcare Limited, Auckland, New Zealand) until SpO2 on pulse oximetry was > 95% and for at least 3 min. A flow of 0.5 l/kg/min-1 was used until induction agents had been administered, and then increased to 2 l/kg/min-1. Nasal oxygenation was continued without ventilation of the lungs while waiting for neuromuscular blockade, and during placing, replacing or repositioning the airway. Anaesthetists were free to carry out bag-mask ventilation of the lungs if they considered this necessary to maintain safe oxygen saturations. After securing the airway, the patient was connected to a circle circuit primed with 100% oxygen and the FIO2 was continued at 100% for a period of at least five more minutes. Relevant times were recorded, including start of pre-oxygenation and start of induction of anaesthesia.
  Arms: high flow nasal oxygen
Procedure: face mask — In the control group, pre-oxygenation was provided using 100% oxygen via a sealed facemask and a circle-absorber anaesthetic circuit primed with 100% oxygen by installing a ventilation bag to the mouthpiece filter and ventilating the circuit with 100% oxygen. Anaesthetists were free to carry out bag-mask ventilation of the lungs once induction medications had been administered.
  Arms: face mask

SUMMARY:
Endotracheal intubation in infants often involves more than one attempt, and oxygen desaturation is common. It is unclear whether nasal high-flow therapy, which extends the time to desaturation during elective intubation in infants receiving general anesthesia, can decrease the occurence of desaturation during intubation.

The investigators tested the hypothesis that high-flow nasal oxygen cannulae would be effective in maintaining oxygen saturation during intubation than facemasks for pre-oxygenation. The investigators randomly allocated 132 patients undergoing elective surgery aged <=12 months to pre-oxygenation using either high-flow nasal oxygen or facemask.

ELIGIBILITY:
Inclusion Criteria:

* Infants undergoing general anesthesia with endotracheal intubation.

Exclusion Criteria:

* infants who diagnosed as cardiorespiratory problem preoperatively.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of oxygen desaturation <95% | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.

SECONDARY OUTCOMES:
Occurrence of oxygen desaturation <90% | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
the lowest oxygen saturation | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
the changes in oxygen reserve index | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
ETCO2 in first breath after intubation | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
ETO2 in first breath after intubation | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
Number of intubation attempts | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
Intubation times | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  time required to securing the airway.
Occurrence of rescue bag mask ventilation | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
Occurrence of gastric insufflation | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Eun-hee Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided